CLINICAL TRIAL: NCT04003974
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, 48-Week, Parallel-Group Study of the Efficacy and Safety of Losmapimod in Treating Subjects With Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Efficacy and Safety of Losmapimod in Subjects With Facioscapulohumeral Muscular Dystrophy (FSHD)
Acronym: FSHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIS-002-2019
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
Keywords: FSHD, FSHD1; Muscular Dystrophies; Muscular Dystrophy; Facioscapulohumeral Muscular Disorders; Musculoskeletal Diseases; Neuromuscular Diseases
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled, 48-week parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed in a double-blind fashion. The investigator, study staff, subjects, sponsor and monitor will remain blinded to the treatment until study closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): FSHD1 patients with genetic confirmation will receive Losmapimod 15 mg twice daily given as two 7.5 mg tablets per dose by mouth; for a total of 4 pills or 30 mg daily for 48 weeks.
  Interventions: Drug: Losmapimod oral tablet
- Placebo (Placebo Comparator): FSHD1 patients with genetic confirmation will receive a Placebo twice daily given as two 7.5 mg tablets per dose by mouth; for a total of 4 pills or 30 mg daily for 48 weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Losmapimod oral tablet — Losmapimod will be administered with food when possible.
  Arms: Treatment
Drug: Placebo oral tablet — Placebo will be administered with food when possible
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety and efficacy of Losmapimod in treating patients with Facioscapulohumeral Muscular Dystrophy (FSHD) over 48 weeks.

DETAILED DESCRIPTION:
This study is a Phase 2, randomized, double-blind, placebo-controlled, parallel-group, multicenter study designed to evaluate the efficacy and safety of losmapimod in treating patients with Facioscapulohumeral Muscular Dystrophy (FSHD) over 48 weeks. Patients will participate in this study for approximately 53 weeks. This will include a 4-week screening period, a 48-week, placebo-controlled treatment period and a 7 day safety follow-up period. Patients must have a confirmed diagnosis of FSHD1 and genetic confirmation must be obtained prior to the screening MRI and baseline muscle biopsy. Patients will be randomized to receive 15 mg of losmapimod or placebo twice daily given as two 7.5 mg tablets per dose by mouth; for a total of 4 pills or 30 mg daily for 48 weeks. All patients will be asked to attend the study clinic for each scheduled visit.

The primary endpoint of the study is to evaluate the efficacy of losmapimod in inhibiting or reducing expression of DUX4, as measured by a subset of DUX4-regulated gene transcripts in skeletal muscle biopsies of FSHD patients. Secondary endpoints include evaluation of the safety and tolerability of losmapimod, the plasma concentrations of losmapimod, levels of losmapimod in skeletal muscle and losmapimod target engagement in blood and skeletal muscle in FSHD patients.

This study was conducted during the Coronavirus Disease-2019 (COVID-19) Pandemic. The pandemic restrictions limited some assessments in the FSHD1 population in the clinic, including collection of some data for Week 24.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have consented to participate and must have provided signed, dated and witnessed IRB-approved informed consent form that conforms to federal and institutional guidelines.
* Male or female subjects
* Confirmed diagnosis of FSHD1 with 1 to 9 repeats via assessment of the size of the D4Z4 array on chromosome 4. Genetic confirmation must be obtained prior to the screening MRI and baseline muscle biopsy.
* Clinical severity score of 2 to 4 (RICCI Score; Range 0-5), inclusive at screening
* Must have a MRI-eligible muscle for biopsy
* Must be willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines and other study procedures.
* Will practice an approved method of birth control

Exclusion Criteria:

* Has a history of any illness or any clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include, but is not limited to, a history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; neuromuscular diseases except FSHD (eg, myopathy, neuropathy, neuromuscular junction disorders); or clinically significant history of mental disease.
* For subjects who are on drug(s) or supplements that may affect muscle function, as determined by the treating physician, or that are included in the list of drugs presented in the protocol, subjects must be on a stable dose of that drug(s) or supplement for at least 3 months prior to the first dose of study drug and remain on that stable dose for the duration of the study. Changes to the dose or treatment discontinuation during the study can only be done for strict medical reasons by the treating physician with clear documentation and notification to the sponsor.
* Acute or chronic history of liver disease or known to have current alanine aminotransferase ≥2 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN, or known history of hepatitis B or C.
* Known severe renal impairment (defined as a glomerular filtration rate of <30 mL/min/1.73m2).
* Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or antibodies against human immunodeficiency virus (HIV)-1 and -2.
* Male subjects with a female partner who is planning to become pregnant during the study or within 90 days after the last dose of study drug.
* Use of another investigational product within 30 days or 5 half-lives (whichever is longer), or according to local regulations, or currently participating in a study with an investigational product. Note: concurrent participation in other non-drug studies may be acceptable if confirmed in writing by the sponsor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Mellion, MD, Study Director — Fulcrum Therapeutics
Locations (17):
- United States (12):
  - University of California Irvine, Irvine, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washinton Medical Center, Seattle, Washington
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- CHU de NICE- CHU pasteur2, Nice, France
- Spain (2):
  - Hospital de la Sta Creu i St Pau, Barcelona
  - Hospital UiP La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- [Background] Cheriyan J, Webb AJ, Sarov-Blat L, Elkhawad M, Wallace SM, Maki-Petaja KM, Collier DJ, Morgan J, Fang Z, Willette RN, Lepore JJ, Cockcroft JR, Sprecher DL, Wilkinson IB. Inhibition of p38 mitogen-activated protein kinase improves nitric oxide-mediated vasodilatation and reduces inflammation in hypercholesterolemia. Circulation. 2011 Feb 8;123(5):515-23. doi: 10.1161/CIRCULATIONAHA.110.971986. Epub 2011 Jan 24. PMID 21262998
- [Background] de Greef JC, Lemmers RJ, van Engelen BG, Sacconi S, Venance SL, Frants RR, Tawil R, van der Maarel SM. Common epigenetic changes of D4Z4 in contraction-dependent and contraction-independent FSHD. Hum Mutat. 2009 Oct;30(10):1449-59. doi: 10.1002/humu.21091. PMID 19728363
- [Background] Han JJ, Kurillo G, Abresch RT, de Bie E, Nicorici A, Bajcsy R. Reachable workspace in facioscapulohumeral muscular dystrophy (FSHD) by Kinect. Muscle Nerve. 2015 Feb;51(2):168-75. doi: 10.1002/mus.24287. Epub 2014 Nov 19. PMID 24828906
- [Background] Jagannathan S, Shadle SC, Resnick R, Snider L, Tawil RN, van der Maarel SM, Bradley RK, Tapscott SJ. Model systems of DUX4 expression recapitulate the transcriptional profile of FSHD cells. Hum Mol Genet. 2016 Oct 15;25(20):4419-4431. doi: 10.1093/hmg/ddw271. PMID 28171552
- [Background] Statland JM, Tawil R. Risk of functional impairment in Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2014 Apr;49(4):520-7. doi: 10.1002/mus.23949. Epub 2014 Feb 10. PMID 23873337
- [Background] Wang LH, Friedman SD, Shaw D, Snider L, Wong CJ, Budech CB, Poliachik SL, Gove NE, Lewis LM, Campbell AE, Lemmers RJFL, Maarel SM, Tapscott SJ, Tawil RN. MRI-informed muscle biopsies correlate MRI with pathology and DUX4 target gene expression in FSHD. Hum Mol Genet. 2019 Feb 1;28(3):476-486. doi: 10.1093/hmg/ddy364. PMID 30312408
- [Derived] Tawil R, Wagner KR, Hamel JI, Leung DG, Statland JM, Wang LH, Genge A, Sacconi S, Lochmuller H, Reyes-Leiva D, Diaz-Manera J, Alonso-Perez J, Muelas N, Vilchez JJ, Pestronk A, Gibson S, Goyal NA, Hayward LJ, Johnson N, LoRusso S, Freimer M, Shieh PB, Subramony SH, van Engelen B, Kools J, Leinhard OD, Widholm P, Morabito C, Moxham CM, Cadavid D, Mellion ML, Odueyungbo A, Tracewell WG, Accorsi A, Ronco L, Gould RJ, Shoskes J, Rojas LA, Jiang JG. Safety and efficacy of losmapimod in facioscapulohumeral muscular dystrophy (ReDUX4): a randomised, double-blind, placebo-controlled phase 2b trial. Lancet Neurol. 2024 May;23(5):477-486. doi: 10.1016/S1474-4422(24)00073-5. PMID 38631764
- [Derived] Jagannathan S, de Greef JC, Hayward LJ, Yokomori K, Gabellini D, Mul K, Sacconi S, Arjomand J, Kinoshita J, Harper SQ. Meeting report: the 2021 FSHD International Research Congress. Skelet Muscle. 2022 Jan 17;12(1):1. doi: 10.1186/s13395-022-00287-8. PMID 35039091

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was a randomized, double-blind placebo-controlled treatment period for 48 weeks which evaluated the efficacy and safety of losmapimod.
Groups:
- Losmapimod 15 Milligrams (mg) Twice Daily (BID): Participants were randomized to receive losmapimod tablets 15 mg (2×7.5 mg tablets/dose BID) orally (PO) for 48 weeks
- Placebo: Participants were randomized to receive matching placebo tablets PO BID for 48 weeks.
Period: Overall Study
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Missing | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: included all participants who were randomly assigned to receive double-blind study drug in the placebo-controlled treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.7 (12.44) | 45.7 (12.69) | 45.7 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 28 | 26 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 37 | 36 | 73
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 39 | 70
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Double Homeobox 4 (DUX4) Activity in Affected Skeletal Muscle
Description: Skeletal muscle biopsies were collected at Baseline and post-Baseline. DUX4 activity in skeletal muscle biopsies was assessed by measuring expression levels of a panel of 6 genes known to be regulated by DUX4. Expression levels of genes were measured using a validated quantitative RT-PCR assay and expressed as Ct (PCR cycles). Raw Ct for each of the 6 genes was normalized to the specified reference genes to generate a normalized Ct. The DUX4 activity is the average of the normalized Cts of each of the identified 6 genes, where the Ct for each of the 6 genes is first normalized to reference genes before the average is generated. Change in Baseline is calculated as [average delta Ct across the 6 genes post-baseline] minus [average delta Ct across the 6 genes at baseline].
Time Frame: Baseline and Week 16 to Week 36
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Delta threshold cycle (Ct)
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 39 | 38
Delta threshold cycle (Ct) | 0.8292 (0.6138) | 0.4008 (0.6491)
Statistical Analysis 1: Comparison: Losmapimod 15 Milligrams (mg) Twice Daily (BID) vs Placebo; Test type: Other — Mean DUX4 activity was derived for each participant at each time point (Baseline and post-Baseline) based on normalized gene expression values for the 6-gene panel. Changes from Baseline to post-Baseline were analyzed using an ANCOVA model; p = 0.5621, ANCOVA; Least square mean difference = 0.4284, 95% CI 2-sided [-1.0376 to 1.8945] — Results are expressed as difference in Least-Squares (LS) means of the changes from Baseline to post-Baseline in DUX4 activity for each group, losmapimod and placebo

2. Secondary Outcome: Number of Participants With Type of Adverse Events (AEs) to Losmapimod
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A Serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. A treatment emergent adverse events (TEAE) is defined as any event that was not present before exposure to study drug or any event that was already present but worsens in either intensity or frequency after exposure to study drug. Number of participants with type of AEs to losmapimod has been presented which included: TEAEs and SAEs.
Time Frame: Up to Week 48
Population: Safety Analysis Set: included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Type: TEAEs | 29 | 23
  Type: SAEs | 2 | 0

3. Secondary Outcome: Number of Participants With Severity of AEs to Losmapimod
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with severity grading of AEs to losmapimod has been presented: Mild (An event that is usually transient in nature and generally does not interfere with normal activities), Moderate (An AE that is sufficiently discomforting to interfere with normal activities) and Severe (An AE that is incapacitating and prevents normal activities). The higher the grade, the more severe the symptoms.
Time Frame: Up to Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Severity: Mild | 18 | 15
  Severity: Moderate | 9 | 8
  Severity: Severe | 2 | 0

4. Secondary Outcome: Number of Participants With Relationship of AEs to Losmapimod
Description: An AE is any untoward medical occurrence in a clinical study participant,temporally associated with use of a study intervention, whether or not considered related to study intervention. An SAE is any untoward medical occurrence that, at any dose results in death,is life-threatening,requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with relationship of AEs to losmapimod has been presented:Unlikely related(most likely produced by other factors and temporal relationship of AE to drug makes a causal relationship unlikely),not related (no association between drug and AE), possibly related (treatment with drug caused/contributed to AE),probably related (reasonable temporal sequence of event with drug exists) and definitely related (definite causal relationship exists between drug and AE)
Time Frame: Up to Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Relationship: Unlikely related | 4 | 7
  Relationship: Not related | 16 | 14
  Relationship: Possibly related | 9 | 1
  Relationship: Probably related | 0 | 1
  Relationship: Definitely related | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) is one of scientific and medical concern for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate. Adverse events of special interest for this study included liver tests that met the criteria for potential drug-induced liver injury (DILI), in accordance with the Unites States (US) Food and Drug Administration (FDA) Guidance for Industry-Drug-Induced Liver Injury: Premarketing Clinical Evaluation. Number of participants with AESIs has been presented.
Time Frame: Up to Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Who Prematurely Discontinued Study Drug Due to a Treatment Emergent Adverse Event (TEAE)
Description: TEAE was an AE that began on or after the first dose of study drug and before the stop of study drug + 7 days or begins before the first dose of study drug and worsened in severity on or after the first dose of study drug and before the stop of study drug + 7 days. An AE with completely missing onset and end dates were considered as treatment-emergent AE. Number of participants who prematurely discontinued study drug due to a TEAE has been presented.
Time Frame: Up to Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

7. Secondary Outcome: Change From Baseline in Muscle Fat Fraction (MFF) at Week 12, Week 24 and Week 48
Description: Measurement of the extent of skeletal muscle tissue replacement by fat in FSHD participants were done through automatic skeletal muscle segmentation for the 3D muscle volumes and fat fraction analysis via robust algorithms using Dixon imaging. Composite variables, incorporating pre-selected muscles, were derived for longitudinal analysis of MFF. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 12, Week 24 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 30 | 29
Percentage point
  Week 12: number analyzed (Participants) | 30 | 26
  Week 12 | 0.53 (1.433) | 0.52 (1.783)
  Week 24: number analyzed (Participants) | 8 | 7
  Week 24 | 0.45 (1.053) | 0.99 (1.723)
  Week 48: number analyzed (Participants) | 24 | 29
  Week 48 | 1.22 (2.269) | 1.67 (2.011)

8. Secondary Outcome: Change From Baseline in Lean Muscle Volume (LMV) at Week 12, Week 24 and Week 48
Description: Measurement of the extent of skeletal muscle tissue replacement by fat in FSHD participants were done through automatic skeletal muscle segmentation for the 3D muscle volumes and fat fraction analysis via robust algorithms using Dixon imaging. Composite variables, incorporating pre-selected muscles, were derived for longitudinal analysis of LMV. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 12, Week 24 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 30 | 29
Liter
  Week 12: number analyzed (Participants) | 30 | 26
  Week 12 | -0.02 (0.069) | -0.01 (0.067)
  Week 24: number analyzed (Participants) | 8 | 7
  Week 24 | 0.00 (0.032) | -0.04 (0.045)
  Week 48: number analyzed (Participants) | 24 | 29
  Week 48 | -0.10 (0.093) | -0.10 (0.114)

9. Secondary Outcome: Change From Baseline in Muscle Fat Infiltration (MFI) at Week 12, Week 24 and Week 48
Description: Measurement of the extent of skeletal muscle tissue replacement by fat in FSHD participants were done through automatic skeletal muscle segmentation for the 3D muscle volumes and fat fraction analysis via robust algorithms using Dixon imaging. Composite variables, incorporating pre-selected muscles, were derived for longitudinal analysis of MFI. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 12, Week 24 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 30 | 29
Percentage point
  Week 12: number analyzed (Participants) | 30 | 26
  Week 12 | -0.02 (0.842) | 0.24 (0.547)
  Week 24: number analyzed (Participants) | 8 | 7
  Week 24 | -0.16 (0.438) | 0.49 (0.921)
  Week 48: number analyzed (Participants) | 24 | 29
  Week 48 | 0.07 (0.796) | 0.47 (0.655)

10. Secondary Outcome: Plasma Concentration After Administration of Losmapimod
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of losmapimod.
Time Frame: Pre dose, 4 hours post dose, Week 4 pre dose, Week 4: 4 hours post dose, Week 12, Week 16 pre dose, Week 16: 4 hours post dose, Week 24, Week 36 pre dose, Week 36: 4 hours post dose, Week 48
Population: Pharmacokinetics Analysis Set: included all participants who received at least 1 dose of losmapimod and had an evaluable PK data for losmapimod. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Nanogram per milliliter
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 40
Nanogram per milliliter
  Pre dose | NA [NA to NA] — NA indicates that Median and full range could not be calculated as the values were Below the level of quantification (BLQ)
  4 hours post dose | 61.200 [6.56 to 147.00]
  Week 4 pre dose: number analyzed (Participants) | 36
  Week 4 pre dose | 27.000 [3.54 to 120.00]
  Week 4: 4 hours post dose: number analyzed (Participants) | 38
  Week 4: 4 hours post dose | 87.600 [46.40 to 165.00]
  Week 12: number analyzed (Participants) | 31
  Week 12 | 58.300 [15.40 to 232.00]
  Week 16 pre dose: number analyzed (Participants) | 25
  Week 16 pre dose | 31.900 [0.10 to 110.00]
  Week 16: 4 hours post dose: number analyzed (Participants) | 26
  Week 16: 4 hours post dose | 82.450 [21.30 to 145.00]
  Week 24: number analyzed (Participants) | 26
  Week 24 | 62.150 [0.10 to 239.00]
  Week 36 pre dose: number analyzed (Participants) | 27
  Week 36 pre dose | 25.100 [0.10 to 77.10]
  Week 36: 4 hours post dose: number analyzed (Participants) | 26
  Week 36: 4 hours post dose | 68.200 [37.60 to 182.00]
  Week 48: number analyzed (Participants) | 28
  Week 48 | 73.400 [0.51 to 163.00]

11. Secondary Outcome: Concentration of Losmapimod in Skeletal Muscle Biopsy
Description: Skeletal muscle biopsy samples were collected at indicated time points for the assessment of concentration of losmapimod.
Time Frame: Baseline, Week 16 and Week 36
Population: Pharmacokinetics Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Nanogram per gram
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID)
Number analyzed (Participants) | 16
Nanogram per gram
  Baseline: number analyzed (Participants) | 10
  Baseline | 0.301 [0.13 to 68.40]
  Week 16 | 56.450 [14.10 to 117.00]
  Week 36: number analyzed (Participants) | 9
  Week 36 | 93.800 [37.30 to 144.00]

12. Secondary Outcome: Percent Change From Baseline in Phosphorylated Heat Shock Protein 27 (pHSP27)/Total Heat Shock Protein 27 (tHSP27)
Description: Blood samples were collected for Pharmacodynamic (PD) analysis of pHSP27/tHSP27. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Percent change from Baseline was defined as value of post Baseline minus Baseline value divided by Baseline value and multiplied by 100.
Time Frame: Baseline and at Day 1: 4 hours post dose, Week 16: pre dose, Week 16: 4 hours post dose, Week 36 pre dose, Week 36: 4 hours post dose
Population: Pharmacodynamics Analysis Set: included all participants who received at least 1 dose of losmapimod and have evaluable PD data for losmapimod. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 35 | 35
Percent change
  Day 1: 4 hours post dose | -34.228 (21.3731) | 10.968 (41.3115)
  Week 16: pre dose: number analyzed (Participants) | 21 | 16
  Week 16: pre dose | 16.392 (102.7915) | 39.497 (92.6947)
  Week 16: 4 hours post dose: number analyzed (Participants) | 22 | 15
  Week 16: 4 hours post dose | -18.888 (59.0971) | 34.176 (83.1994)
  Week 36 pre dose: number analyzed (Participants) | 16 | 22
  Week 36 pre dose | -46.203 (28.4928) | 20.445 (203.8013)
  Week 36: 4 hours post dose: number analyzed (Participants) | 17 | 21
  Week 36: 4 hours post dose | -62.250 (18.6709) | -8.908 (74.6476)

13. Other Pre Specified Outcome: Change From Baseline in Reachable Work Space (RWS) Dominant and Non-dominant Total Relative Surface Area (RSA) With Weight Quintant (Q)1 to Q5
Description: The RWS was a 3-dimensional sensor-based system (using a single depth-ranging sensor) that could unobtrusively detect an individual's RWS and reflect an individual global upper extremity function, including shoulder and proximal arm. Participants were seated in front of a 3D camera and asked to perform a standardized upper extremity movement protocol under the supervision of a study clinical evaluator with and without weights and on both the right and left arms at indicated time points. The absolute total RWS surface envelope area as well as areas for each of the quadrants was calculated and provided in a blinded fashion, with no access to treatment assignment information. The RWS RSA represented the portion of the unit hemisphere that was covered by an individual's hand movement. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 37 | 39
Unitless
  Week 4: Dominant Total RSA Weighted Q1 to Q5 | -0.0009 (0.07652) | -0.0022 (0.06615)
  Week 12: Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 28 | 25
  Week 12: Dominant Total RSA Weighted Q1 to Q5 | 0.0109 (0.09214) | -0.0069 (0.09547)
  Week 24: Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 24 | 27
  Week 24: Dominant Total RSA Weighted Q1 to Q5 | -0.0066 (0.10246) | -0.0094 (0.10672)
  Week 36: Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 25 | 29
  Week 36: Dominant Total RSA Weighted Q1 to Q5 | -0.0169 (0.09346) | -0.0371 (0.12235)
  Week 48: Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 25 | 28
  Week 48: Dominant Total RSA Weighted Q1 to Q5 | 0.0103 (0.07273) | -0.0267 (0.08972)
  Week 4: Non-Dominant Total RSA Weighted Q1 to Q5 | 0.0077 (0.07212) | 0.0189 (0.07697)
  Week 12: Non-Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 29 | 25
  Week 12: Non-Dominant Total RSA Weighted Q1 to Q5 | 0.0156 (0.07221) | 0.0084 (0.08577)
  Week 24: Non-Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 24 | 27
  Week 24: Non-Dominant Total RSA Weighted Q1 to Q5 | 0.0259 (0.06960) | 0.0114 (0.09087)
  Week 36: Non-Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 25 | 29
  Week 36: Non-Dominant Total RSA Weighted Q1 to Q5 | 0.0287 (0.09934) | -0.0069 (0.09770)
  Week 48: Non-Dominant Total RSA Weighted Q1 to Q5: number analyzed (Participants) | 25 | 29
  Week 48: Non-Dominant Total RSA Weighted Q1 to Q5 | 0.0169 (0.09090) | -0.0129 (0.09841)

14. Other Pre Specified Outcome: Change From Baseline in Classic Timed Up and Go (TUG) Average Completion Time
Description: The TUG test was a simple test that was used to assess a person's mobility and required both static and dynamic balance. It measured the time that a person takes to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The optimized TUG test was the classic TUG but added the component of getting up from a laying position on a bed-like table in the clinic at the start of the test and laying back down on his or her back at the end of the test. Participants were timed as they started from a seated or laying position, rise to a standing position, walked a total of 6 meters and then returned to either a seated or laying position. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value
Time Frame: Baseline and at Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 39 | 39
Seconds
  Week 4 | 2.011 (16.8603) | 0.297 (2.0577)
  Week 12: number analyzed (Participants) | 30 | 25
  Week 12 | -0.340 (2.5908) | 0.183 (1.7839)
  Week 24: number analyzed (Participants) | 23 | 26
  Week 24 | 0.960 (2.8012) | 0.384 (1.9678)
  Week 36: number analyzed (Participants) | 25 | 30
  Week 36 | 0.252 (2.8725) | 0.709 (1.6041)
  Week 48: number analyzed (Participants) | 25 | 29
  Week 48 | -0.340 (2.1289) | 0.789 (1.7059)

15. Other Pre Specified Outcome: Change From Baseline in Facioscapulohumeral Muscular Dystrophy (FSDH) TUG Average Completion Time
Description: as for outcome 14
Time Frame: Baseline and at Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 36 | 38
Seconds
  Week 4 | -0.993 (3.4234) | 0.750 (2.1824)
  Week 12: number analyzed (Participants) | 29 | 25
  Week 12 | -0.380 (2.7827) | 0.058 (1.7805)
  Week 24: number analyzed (Participants) | 23 | 26
  Week 24 | 0.549 (2.9794) | 0.304 (1.8555)
  Week 36: number analyzed (Participants) | 24 | 29
  Week 36 | -0.653 (4.1121) | 0.389 (1.7394)
  Week 48: number analyzed (Participants) | 23 | 30
  Week 48 | 0.342 (3.7028) | 0.334 (2.0296)

16. Other Pre Specified Outcome: Change From Baseline in All Muscles Total Average Strength as Assessed by Hand-held Dynamometry
Description: Quantitative isometric dynamometry (hand-held dynamometer) was used to assess the skeletal muscles strength of study participants in both the upper and lower limbs bilaterally. The MicroFET2 hand-held dynamometer was used to measure strength in the bilateral shoulders, elbow flexors and extensors, and ankle dorsiflexors. The Jamar Plus Digital Hand Dynamometer was used to measure bilateral grip strengths. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 4, Week 12, Week 24, Week 36 and Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 38 | 39
Kilograms
  Week 4 | 5.064 (15.3103) | -1.386 (9.2043)
  Week 12: number analyzed (Participants) | 29 | 25
  Week 12 | 1.439 (11.5791) | -0.230 (9.5417)
  Week 24: number analyzed (Participants) | 24 | 26
  Week 24 | -1.551 (22.8920) | -9.477 (15.6318)
  Week 36: number analyzed (Participants) | 25 | 30
  Week 36 | -3.608 (33.1467) | -11.772 (22.7106)
  Week 48: number analyzed (Participants) | 25 | 30
  Week 48 | -5.358 (22.0734) | -15.021 (28.3042)

17. Other Pre Specified Outcome: Change From Baseline in Motor Function Measure (MFM) Domain 1 Score
Description: The MFM scale assessed the severity of the motor deficit as determined by an experienced physical therapist. The MFM domain 1 was a validated evaluator administered functional measure for neuromuscular disorders, with 13 items related to standing and transfers. Generic Values for each domain were: 0 = cannot perform the task, 1 = initiated the task, 2 - performs the movement incompletely, or completely but imperfectly, 3 = performs the task fully and 'normally'. Total score was the sum of all the domains for D1 divided by the maximum score possible and multiplied by 100. Min=0, Max = 100. Lower numbers on the scale represented a worse outcome. Baseline was defined as the last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 25 | 30
Scores on a scale | 2.76 (9.079) | 2.00 (8.780)

18. Other Pre Specified Outcome: Change From Baseline in FSHD Health Index (HI)
Description: The FSHD-HI was a 15-domain questionnaire designed and based on participant interviews to measure total FSHD health-related quality-of-life, including both motor impairment and the social and emotional impact of FSHD. 116 questions were combined into a total score, the score is transformed onto a percentage scale, with score ranging from 0 (no disability) to 100 (maximal disability); lower scores represented decreasing disability. Baseline was defined as last non-missing evaluation on or before the day of first dose of study drug. Change from Baseline was calculated as Baseline minus post-dose value.
Time Frame: Baseline and at Week 48
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 28 | 30
Scores on a scale | 1.17 (13.499) | -0.64 (8.024)

19. Other Pre Specified Outcome: Number of Participants With Improved and Not Improved Response to Patients' Global Impression of Change (PGIC)
Description: The PGI-C was a one-time assessment to measure the participant's impression of the how their illness had changed over time. It is a single question that assessed on a scale of 1-7 if there has been an improvement, decline or no change in clinical status. The score ranged from: Responses of 1= Very much improved, 2= Much improved, and 3= Minimally improved which were considered as improved and responses of 4 = No change, 5 = Minimally worse, 6= Much worse, and 7=Very much worse were considered as not improved. Higher scores indicated worse symptoms.
Time Frame: At Week 48
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Improved: Week 48 | 8 | 2
  Not Improved: Week 48 | 21 | 29

ADVERSE EVENTS:
Time Frame: Up to Week 48
Description: Safety population which included all participants who received any study drug.
Arm/Group | Losmapimod 15 Milligrams (mg) Twice Daily (BID) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40 | 0/40
Other Adverse Events (participants affected / at risk) | 29/40 | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=40) | Placebo (N=40)
Postoperative wound infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losmapimod 15 Milligrams (mg) Twice Daily (BID) (N=40) | Placebo (N=40)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 6 | 2
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Incision site rash (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dental necrosis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 5
Hypoaesthesia (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 1 | 0
Postural tremor (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood iron decreased (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Erythema of eyelid (Eye disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT04003974/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT04003974/SAP_001.pdf